CLINICAL TRIAL: NCT07313852
Title: A Phase II Study of Concurrent Inotuzumab and Subcutaneous Blinatumomab in Older or Unfit Adult Patients With Newly Diagnosed B-cell Acute Lymphoblastic Leukemia
Brief Title: A Study of Inotuzumab and Blinatumomab in People With Newly Diagnosed B-cell Acute Lymphoblastic Leukemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26-035
Record Dates: First submitted 2025-12-30; First posted 2026-01-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; B-Cell Acute Lymphoblastic Leukemia, Adult; B-ALL
Keywords: B-cell Acute Lymphoblastic Leukemia; B-Cell Acute Lymphoblastic Leukemia, Adult; B-ALL; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Burkitt Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants With Newly Diagnosed B-cell Acute Lymphoblastic Leukemia (Experimental): Participants will be newly diagnosed with CD19+ and CD22+ B-cell Acute Lymphoblastic Leukemia
  Interventions: Drug: Blinatumomab Injection

INTERVENTIONS:
Drug: Blinatumomab Injection — Blinatumomab given via subcutaneous injection

SUMMARY:
The purpose of this study is to find out whether combining inotuzumab and blinatumomab is a safe and effective treatment for participants with newly diagnosed B-cell acute lymphoblastic leukemia (B-ALL).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age.
* Newly diagnosed CD19+ and CD22+ B-ALL.

  * Patients ≥55 years old, OR
  * Patients 18-54 years old who decline or are deemed unfit for conventional chemotherapy with at least one of the following critieria:
* ECOG performance status of 2 or more
* Severe cardiac comorbidity (including congestive heart failure requiring treatment, ejection fraction ≤50% but greater than 40%)
* Known pulmonary comorbidity (including DLCO ≤65% or FEV1 ≤65%)
* Renal comorbidity (including creatinine clearance 30-70 mL/min)
* Any other comorbidity that the physician judges to be incompatiable with chemotherapy
* Patients with isolated extramedullary disease will be allowed as long as they have identifiable disease by PET CT at time of enrollment.
* Philadelphia chromosome negative by FISH/karyotype for t(19;22) or RT PCR for bcr-abl transcript.
* CD19 and CD22 expression will be confirmed by enrolling institutions prior to study registration by flow cytometry and/or IHC.
* Creatinine ≤2.0 mg/100 ml or creatinine clearance ≥30 mL/min
* Direct bilirubin ≤2.0 mg/100 ml, AST and ALT ≤3.0x upper limit of normal (ULN)

Exclusion Criteria:

* Patients with Burkitt's lymphoma, T-ALL, CML in lymphoid blast crisis and mixed phenotype acute leukemia (MPAL).
* Patients with B-ALL who received prior treatments, with the exception of corticosteroid, hydroxyurea, or one dose of vincristine, are ineligible.
* Patients with Ph+ B-ALL by FISH or RT PCR.
* ECOG performance status >2.
* Left ventricular ejection fraction (LVEF) <40%.
* History of sinusoidal obstruction syndrome (SOS), also known as veno-occlusive disease (VOD).
* Ongoing need for systemic T-cell suppressive therapy (e.g. corticosteroids, tacrolimus, cyclosporine, etc.) for active autoimmune disease or prior solid organ transplantation.
* Pregnant or lactating women. Women and men of childbearing age should use effective contraception while on this study and continue for 1 year after all treatment is finished.
* Patients with HIV or active hepatitis B or hepatitis C infection are ineligible.
* Patients with concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation or hormonal therapy, with the exception of squamous and basal cell carcinoma of the skin, in situ cervical cancer, adequately treated stage I/II cancer from which the patient is current in complete remission, or any other cancer from which the patient has been disease free for five years
* Patients with history or presence of clinically significant neurological disorders such as epilepsy, generalized seizure disorder, or severe brain injuries.
* Any other issue which, in the opinion of the treating physician, would make the patient ineligible for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Rate of MRD negative CR/CRi at the end of induction | up to 1 year
  To evaluate the efficacy of concurrent inotuzumab and subcutaneous blinatumomab in patients older (≥55) or 18-55 years that refuse or are unfit for intensive chemotherapy with newly diagnosed B-cell Acute Lymphoblastic Leukemia as assessed by rate of MRD negative CR/CRi (10-4 threshold) at the end of induction.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org